CLINICAL TRIAL: NCT07124377
Title: Phenotypic Manifestations of Hereditary ATTR Amyloidosis Val50Met Variant in a Non-endemic Area. Descriptive Study
Brief Title: Phenotypic Manifestations of Hereditary ATTR Amyloidosis
Status: Enrolling by invitation | Type: Observational
Sponsor: Hospital 9 de Julio de Las Breñas (Other Government)
Collaborators: Instituto de Cardiología de Corrientes (Other)
Responsible Party: Principal Investigator, Mauricio Tomei, Principal Investigator, Hospital 9 de Julio de Las Breñas
Other Study IDs: hATTR Chaco Cluster
Record Dates: First submitted 2025-08-01; First posted 2025-08-15 (Actual); Last update posted 2025-08-15 (Actual); Status verified 2025-08

CONDITIONS: Hereditary Amyloidosis, Transthyretin-Related
Keywords: hATTR; Non Endemic Area
MeSH Terms: conditions — Amyloidosis, Hereditary, Transthyretin-Related | interventions — Weights and Measures; Temperature; Proprioception; Electrocardiography; Electrocardiography, Ambulatory; Echocardiography, Doppler, Color; Surveys and Questionnaires; Electromyography

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Year
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Carriers of the Val50Met variant: Patients with positive genetic test for patogenic variant of the TTR gene
  Interventions: Other: A complete physical examination of all body systems, including height and body weight; Other: Neurological examination includes motor strength testing; sensory testing with pinprick, light touch, temperature, and proprioception; deep tendon reflexes; and gait assessment.; Diagnostic Test: Electrocardiogram (12-lead ECG); Diagnostic Test: 24-Hour Holter Monitoring; Diagnostic Test: Color Doppler echocardiography with "two-dimensional strain" (longitudinal strain); Other: The Norfolk Quality of Life-Diabetic Neuropathy (QOL-DN); Other: questionnaire, the NIS-LL (Neuropathy Impairment Score in the Lower Limbs); Other: COMPASS-31 (Composite Autonomic Symptom Score-31); Diagnostic Test: Electromyogram (EMG); Diagnostic Test: [99mTc]Tc-DPD scintigraphy; Diagnostic Test: Laboratory assessments

INTERVENTIONS:
Other: A complete physical examination of all body systems, including height and body weight — These interventions will be carried out in a time-controlled population within a family cluster of VAL50MET
Other: Neurological examination includes motor strength testing; sensory testing with pinprick, light touch, temperature, and proprioception; deep tendon reflexes; and gait assessment. — These interventions will be carried out in a time-controlled population within a family cluster of VAL50MET
Diagnostic Test: Electrocardiogram (12-lead ECG) — These interventions will be carried out in a time-controlled population within a family cluster of VAL50MET
Diagnostic Test: 24-Hour Holter Monitoring — These interventions will be carried out in a time-controlled population within a family cluster of VAL50MET
Diagnostic Test: Color Doppler echocardiography with "two-dimensional strain" (longitudinal strain) — These interventions will be carried out in a time-controlled population within a family cluster of VAL50MET
Other: The Norfolk Quality of Life-Diabetic Neuropathy (QOL-DN) — These interventions will be carried out in a time-controlled population within a family cluster of VAL50MET
Other: questionnaire, the NIS-LL (Neuropathy Impairment Score in the Lower Limbs) — These interventions will be carried out in a time-controlled population within a family cluster of VAL50MET
Other: COMPASS-31 (Composite Autonomic Symptom Score-31) — These interventions will be carried out in a time-controlled population within a family cluster of VAL50MET
Diagnostic Test: Electromyogram (EMG) — These interventions will be carried out in a time-controlled population within a family cluster of VAL50MET
Diagnostic Test: [99mTc]Tc-DPD scintigraphy — These interventions will be carried out in a time-controlled population within a family cluster of VAL50MET
Diagnostic Test: Laboratory assessments — Laboratory assessments include blood and urine sample collection for serum chemistry, hematology, and urinalysis, with specific biomarker analyses (troponin T, NT-proBNP, Kappa, and Lambda light chains

SUMMARY:
This study focuses on hereditary transthyretin amyloidosis (ATTRv) with the Val50Met variant in a non endemic aerea

DETAILED DESCRIPTION:
We aim to describe the phenotypic variables including preclinical, cardiological, neurological, and mixed manifestations in patients carrying the Val50Met variant. Our goal is to identify early disease onset criteria in initially asymptomatic patients, enhancing early detection and treatment strategies. Participants will undergo various clinical examinations and tests to gather comprehensive data.

ELIGIBILITY:
Inclusion Criteria:

* All subjects between 20 and 70 years of age, carriers of the Val50Met variant

Exclusion Criteria:

* Patients who refuse to participate.

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All subjects between 20 and 70 years of age, carriers of the Val50Met variant from August 1st ,2024 to December 30st, 2025, belonging to a cluster of hereditary Transthyretin Amyloidosis will be included
Sampling Method: Non-Probability Sample
Enrollment: 57 (Estimated)
Dates: Start 2024-09-01 (Actual); Primary Completion 2025-12-30 (Estimated); Study Completion 2026-03-01 (Estimated)

PRIMARY OUTCOMES:
Describe the phenotypic variables (preclinical, cardiological, neurological and mixed) in patients carrying the TTR Val50Met variant in a non-endemic population. | 2 years
  The predominantly cardiac phenotype includes patients with abnormal ECG due to rhythm disturbance, heart failure, or dyspnea, minimal neurologic or GI symptoms, and diagnostic findings such as interventricular septum hypertrophy (>12 mm), Holter monitoring, and [99mTc]Tc-DPD scintigraphy (Peugerini Score 1-3).
  The predominantly neurologic phenotype features patients with ongoing neurologic or GI symptoms definitively linked to ATTR amyloidosis, without abnormal ECG findings. Key assessments include autonomic neuropathy (orthostatic hypotension, sexual dysfunction), EMG, Norfolk QoL-DN (-4-246), COMPASS-31 (0-100), and NIS-LL (0-88).
  The mixed phenotype includes patients with abnormal ECG and neurologic or GI symptoms of any severity, failing to meet criteria for predominantly cardiac or neurologic phenotypes.

SECONDARY OUTCOMES:
Explore minimum criteria considered for the onset of disease in patients carrying the Val50Met variant initially identified as asymptomatic. | 2 years
  Minimum criteria for disease onset include: (1) one quantified symptom or sign definitively related to the disease, such as sensorimotor neuropathy, autonomic neuropathy, cardiac involvement, or renal/ocular involvement; (2) any symptom probably related with one abnormal test finding; or (3) absence of symptoms with two abnormal test findings.

CONTACTS AND LOCATIONS:
Overall Officials: Mauricio MT Tomei, MD, Principal Investigator — Hospital 9 de Julio de Las Breñas
Locations (1):
- Hospital las Breñas 9 de Julio, Charata, Chaco Province, Argentina

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Saez MS, Aguirre MA, Perez de Arenaza D, Sorroche P, Nucifora E, Posadas Martinez ML. Epidemiology of variant transthyretin amyloidosis at a reference center in Argentina. Mol Genet Genomic Med. 2021 Nov;9(11):e1812. doi: 10.1002/mgg3.1812. Epub 2021 Oct 20. PMID 34668655
- [Background] Conceicao I, Damy T, Romero M, Galan L, Attarian S, Luigetti M, Sadeh M, Sarafov S, Tournev I, Ueda M. Early diagnosis of ATTR amyloidosis through targeted follow-up of identified carriers of TTR gene mutations. Amyloid. 2019 Mar;26(1):3-9. doi: 10.1080/13506129.2018.1556156. Epub 2019 Feb 22. PMID 30793974
- [Background] Maurer MS, Bokhari S, Damy T, Dorbala S, Drachman BM, Fontana M, Grogan M, Kristen AV, Lousada I, Nativi-Nicolau J, Cristina Quarta C, Rapezzi C, Ruberg FL, Witteles R, Merlini G. Expert Consensus Recommendations for the Suspicion and Diagnosis of Transthyretin Cardiac Amyloidosis. Circ Heart Fail. 2019 Sep;12(9):e006075. doi: 10.1161/CIRCHEARTFAILURE.119.006075. Epub 2019 Sep 4. PMID 31480867
- [Background] Gentile L, Coelho T, Dispenzieri A, Conceicao I, Waddington-Cruz M, Kristen A, Wixner J, Diemberger I, Gonzalez-Moreno J, Cariou E, Maurer MS, Plante-Bordeneuve V, Garcia-Pavia P, Tournev I, Gonzalez-Costello J, Duarte AG, Grogan M, Mazzeo A, Chapman D, Gupta P, Glass O, Amass L; THAOS investigators. A 15-year consolidated overview of data in over 6000 patients from the Transthyretin Amyloidosis Outcomes Survey (THAOS). Orphanet J Rare Dis. 2023 Nov 10;18(1):350. doi: 10.1186/s13023-023-02962-5. PMID 37946256